CLINICAL TRIAL: NCT06129656
Title: Cardiac Amyloidosis Registry of University Hospital Leipzig
Status: Recruiting | Type: Observational
Sponsor: University of Leipzig (Other)
Responsible Party: Sponsor
Other Study IDs: UKL_CA_registry
Record Dates: First submitted 2023-10-19; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-10

CONDITIONS: Cardiac Amyloidosis
Keywords: heart failure; cardiac amyloidosis; restrictive cardiomyopathy
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Heart Failure; Cardiomyopathy, Restrictive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac Amyloidosis: Patients with diagnosed cardiac amyloidosis being treated at Leipzig University Hospital.
  Interventions: Other: Routine diagnostics; Other: Routine treatment

INTERVENTIONS:
Other: Routine diagnostics — Data collection of routine diagnostics
Other: Routine treatment — Data collection of routine treatment

SUMMARY:
This is a clinical registry of patients with cardiac amyloidosis being treated at University Hospital Leipzig. The aim of the registry is to collect detailed information about clinical events, symptoms, imaging, biomarkers, comorbidities, and treatment from routine patient management which would not be provided by randomized clinical trails.

DETAILED DESCRIPTION:
Cardiac amyloidosis is increasingly diagnosed since awareness of the disease and therapeutic options increase. There is evidence from clinical trials about warning signs ("red flags"), diagnostic algorithms, and evidence for specific treatment. However, patients in randomized clinical studies are highly selected and do not necessarily reflect clinical practise. Furthermore, large clinical trials do not account for national medical care differences nor provide data about long-term outcome and the associations with comorbidities.

Clinical registries may reflect broad clinical practise and help to characterize cardiac amyloidosis in terms of epidemiology, application of diagnostic methods, the impact of comorbidities, and real-world clinical course. Furthermore, clinical registry studies may validate data from randomized clinical trials, provide information on implementation of treatment, the quality of interventions, monitoring patients during treatment, and inform about the safety of procedures.

The cardiac amyloidosis registry aims to collect data from the routine clinical management of patients with cardiac amyloidosis at the tertiary care University Hospital Leipzig. In particular, obtaining data about clinical events of heart disease, hemodynamic measures from echocardiography and circulation biomarkers, cardiac morphology from different imaging methods, clinical status, functional capacity, quality of life, and impact of comorbidities during the course of the disease will be the goal of this registry.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed cardiac amyloidosis according to current standards

Exclusion Criteria:

* refusal to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with confirmed cardiac amyloidosis who are beeing treated at Department of Cardiology at University Hospital Leipzig.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2033-05 (Estimated); Study Completion 2033-05 (Estimated)

PRIMARY OUTCOMES:
All-cause and cardiac mortality | 10 years
  Mortality
Cumulative rate of patients with worsening heart failure | 10 years
  Heart failure endpoint
Rate of any hospitalizations | 10 years
  Record of any clinical events requiring hospitalization
Change in left ventricular ejection fraction | Every 6-12 months over 10 years
  Change in LVEF assessed by echocardiography or cardiac MRI
Change in left ventricular wall thickness | Every 6-12 months over 10 years
  Change in left ventricular wall thickness/ mass assessed by echocardiography or cardiac MRI
Change in systolic arterial pressure | Every 6-12 months over 10 years
  Change in sPAP assessed by echocardiography
Change in T1 values | Approx. every 12 months over 10 years
  Change in T1 values assessed by cardiac MRI
Change in extracellular volume values | Approx. every 12 months over 10 years
  Change in ECV assessed by cardiac MRI
Change in N-Terminal Pro-B-Type Natriuretic Peptide over time | Every 3-6 months over 10 years
  Change in serum concentration of NT-proBNP
Change in high-sensitivity cardiac troponin T over time | Every 3-6 months over 10 years
  Change in serum concentration of hs-cTnT
Changes in medical treatment for heart failure | Every 3-6 months over 10 years
  Changes in heart failure medication (i.e. diuretics, beta-blocker, renin-angiotensin system inhibitors, mineralocorticoid receptor antagonists, sodium glucose cotransporter type 2 inhibitors) as well as specific treatment for amyloidosis (e.g. tafamidis) is recorded.

SECONDARY OUTCOMES:
Prevalence and incidence of cardiac and non-cardiac comorbidities | Every 3-6 months over 10 years
  Medical history and reports regarding any comorbidities and previous treatment will be assessed in detail at inclusion. Patients are asked for new comorbidities and new treatments at every visit.
New York Heart Association (NYHA) class over time | Every 3-6 months over 10 years
  As parameter of clinical status
Functional capacity over time | Every 3-6 months over 10 years
  Measured using 6 minute walk test
Quality of life over time | Every 3-6 months over 10 years
  Measured via questionnaire (e.g. KCCQ)
Vital signs over time | Every 3-6 months over 10 years
  Blood pressure
Clinical signs of congestion over time | Every 3-6 months over 10 years
  E.g. edema, jugular venous distension, crackles on lung auscultation
Number of cardiovascular interventions | Monitoring continuously over 10 years
  Indication, efficacy and safety of any cardiovascular intervention will be recorded, such as rate of pacemaker implantations, numbers of valve procedures (aortic valve implantation, mitral or tricuspid valve clipping), left atrial appendage occluder implantation, electrophysiological studies and ablation procedures

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Lavall, MD, Principal Investigator — University of Leipzig
Locations (1):
- University Hospital Leipzig, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No